CLINICAL TRIAL: NCT04134949
Title: Effectiveness of Mindfulness Based Cognitive Therapy (MBCT) on for Insomnia and Mental Health of Prisoners
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, Associate Professor, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.QUMS.REC.1397.294
Record Dates: First submitted 2019-10-19; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT (Experimental): consists of eight weekly treatment sessions of 45 to 60 minutes.
  Interventions: Behavioral: Cognitive Behavior Therapy
- MCBT (Experimental): consists of eight weekly treatment sessions of 45 to 60 minutes.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — consists of eight weekly treatment sessions of 45 to 60 minutes.
  Arms: CBT
Behavioral: Mindfulness-Based Cognitive Therapy — consists of eight weekly treatment sessions of 45 to 60 minutes.
  Arms: MCBT

SUMMARY:
Insomnia is highly prevalent in prisoners and is a risk factor for poor mental well-being, depression, suicidality and aggression, all common concerns in this vulnerable population. Improving sleep management options in prison offers the potential to impact positively on a number of these common risk factors. The study aim is to asses psychological intervention for insomnia in prisons.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age
* Clinical level of Insomnia (more than 10 on ISI)
* Meets criteria for Insomnia according to DSM-5 Insomnia Disorder
* Can speak, understand, and write in Persian
* Male

Exclusion Criteria:

* Currently receiving psychological treatment for Insomnia
* presence of a rapidly progressing neurological or medical disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-10-25 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
sleep hygiene behavior | changes in sleep hygiene behavior baseline , 1 month and 6 months follow-up
  A self reported measure will be used with three items to measure how many days the participants had good sleep hygiene behavior.
Sleep Quality | changes in sleep quality baseline , 1 month and 6 months follow-up
  The Pittsburgh Sleep Quality Index includes seven components of subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, the use of sleep medications and day time dysfunctions provide a total score of these seven components that allows us to better understand the quality and quantity of one's sleep. The Pittsburgh Sleep Quality Index is a self-reporting instrument consisting of nine questions designed to measure the quality of sleep disorders in a period of one month. The scale scores range from 0 to 21, with higher scores indicating poor quality of sleep and scores less than 5 considered as high quality of sleep
Insomnia Severity Index | changes in insomnia baseline , 1 month and 6 months follow-up
  The Insomnia Severity Index is a 7-item questionnaire designed to identify cases of insomnia and evaluate treatment outcomes. The Insomnia Severity Index assesses severity of sleep onset, sleep maintenance and early wakening problems, sleep dissatisfaction, and perceived distress caused by sleep problems. It was found to be a clinically useful tool in assessing changes in insomnia symptoms in insomnia treatment research.Higher scores reflecting more severe sleep problems
Sleep Logs | changes in Sleep Logs , 1 month and 6 months follow-up
  Sleep logs provide self-reported subjective sleep, combining self-reports of: latency, total sleep time, and number and frequency of awakenings.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | changes in HADS, 1 month and 6 months follow-up
  Hospital Anxiety and Depression Scale (HADS) questionnaire. The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.
Perceived Stress Scale (PSS) | changes in PSS, 1 month and 6 months follow-up
  The Perceived Stress Scale is the most widely used measure of global perceived stress, and is a robust predictor of health and disease. The Perceived Stress Scale can range from 0 to 40 with higher scores indicating higher perceived stress.
Mindful Attention Awareness Scale | changes in MAAS, 1 month and 6 months follow-up
  The trait Mindful Attention Awareness Scale is a 15-item scale designed to assess a core characteristic of mindfulness. Higher scores on the Mindful Attention Awareness Scale are associated with fewer & less intense current unpleasant & negative emotional states.
psychological well-being | changes in GHQ-12, 1 month and 6 months follow-up
  The General Health Questionnaire (GHQ-12) is a self-administered questionnaire to screen and detect individuals with a diagnosable psychiatric disorder. The higher the General Health Questionnaire scores, the greater the degree to which the subject may suffer from a psychiatric distress

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Qazvin University of Medical Sciences, Qazvin
  - Social Determinants of Health Research Center, Qazvin

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF